CLINICAL TRIAL: NCT04477824
Title: Is Acute Appendicitis Still a Clinical Diagnosis? Use of Preoperative Diagnostic Imaging Before Appendectomy in Denmark During 2000-15.
Brief Title: Is Acute Appendicitis Still a Clinical Diagnosis?
Status: Completed | Type: Observational
Sponsor: Claus Anders Bertelsen, PhD, MD (Other)
Responsible Party: Sponsor-Investigator, Claus Anders Bertelsen, PhD, MD, Associate professor, consultant surgeon, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Other Study IDs: APP-DIM
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Appendicitis
Keywords: Appendicitis; Appendectomy; Preoperative diagnostic imaging
MeSH Terms: conditions — Appendicitis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic imaging — Ultrasonography, computerized tomography, magnetic resonance imaging

SUMMARY:
This study aims to investigate the use of preoperative diagnostic imaging before appendectomy in Denmark and whether it has changed over time during the period from 2000-15. Secondly, the study aims to investigate regional, age and gender differences in the same setting.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of abdominal pain (1) and appendectomy is the most common emergency surgical procedure performed worldwide (2). During the last decades, there has been a paradigm shift in both diagnosis and treatment of appendicitis - surgical treatment has changed from open to laparoscopic appendectomy (3). Acute appendicitis has traditionally been a clinical diagnosis, but the use of preoperative diagnostic imaging has, in some countries, increased dramatically (4). The use of computed tomography (CT) before appendectomy is in the United States up to 90%, in England 13% and in Holland almost all patients undergo ultrasound and/or CT before appendectomy (1).

The use of antibiotics can be successful in the treatment of uncomplicated appendicitis verified on CT, and the use of CT has significantly lowered the negative appendectomy rate compared to clinical evaluation only (1). But the use of CT is inevitably inducing radiation and increasing lifetime risk of cancer - especially in younger patients who most frequently present with acute appendicitis (1,5). It is estimated that CT of the abdominal region can avoid 12 negative appendectomies but at the cost of one cancer death due to radiation (5). In Denmark surgery is still the only treatment for appendicitis, but how is appendicitis diagnosed? Is acute appendicitis still a clinical diagnosis?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis for appendicitis undergoing appendectomy during the same admission during the period 2000-15

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Denmark with a diagnosis for appendicitis undergoing appendectomy during the same admission during the period 2000-15
Sampling Method: Non-Probability Sample
Enrollment: 82000 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Annual percentage use diagnostic imaging before appendectomy | 24 hours
  Annual percentage use of abdominal ultrasonography, abdominal computerized tomography (with or without contrast) and abdominal MRI 24 hours before appendectomy for appendicitis.

SECONDARY OUTCOMES:
Differences in use of ultrasonography. | 24 hours
  Differences in use of ultrasonography between gender, age groups divided into decades and the five Danish administrative regions.
Differences in use of abdominal computerized tomography (with or without contrast) | 24 hours
  Differences in use of abdominal computerized tomography (with or without contrast) between gender, age groups divided into decades and the five Danish administrative regions.
Differences in use of magnetic resonance imaging | 24 hours
  Differences in use of magnetic resonance imaging between gender, age groups divided into decades and the five Danish administrative regions.

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, Phd, Study Chair — Nordsjaellands Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rud B, Vejborg TS, Rappeport ED, Reitsma JB, Wille-Jorgensen P. Computed tomography for diagnosis of acute appendicitis in adults. Cochrane Database Syst Rev. 2019 Nov 19;2019(11):CD009977. doi: 10.1002/14651858.CD009977.pub2. PMID 31743429
- [Background] GlobalSurg Collaborative. Mortality of emergency abdominal surgery in high-, middle- and low-income countries. Br J Surg. 2016 Jul;103(8):971-988. doi: 10.1002/bjs.10151. Epub 2016 May 4. PMID 27145169
- [Background] Di Saverio S, Birindelli A, Kelly MD, Catena F, Weber DG, Sartelli M, Sugrue M, De Moya M, Gomes CA, Bhangu A, Agresta F, Moore EE, Soreide K, Griffiths E, De Castro S, Kashuk J, Kluger Y, Leppaniemi A, Ansaloni L, Andersson M, Coccolini F, Coimbra R, Gurusamy KS, Campanile FC, Biffl W, Chiara O, Moore F, Peitzman AB, Fraga GP, Costa D, Maier RV, Rizoli S, Balogh ZJ, Bendinelli C, Cirocchi R, Tonini V, Piccinini A, Tugnoli G, Jovine E, Persiani R, Biondi A, Scalea T, Stahel P, Ivatury R, Velmahos G, Andersson R. WSES Jerusalem guidelines for diagnosis and treatment of acute appendicitis. World J Emerg Surg. 2016 Jul 18;11:34. doi: 10.1186/s13017-016-0090-5. eCollection 2016. PMID 27437029
- [Background] Raja AS, Wright C, Sodickson AD, Zane RD, Schiff GD, Hanson R, Baeyens PF, Khorasani R. Negative appendectomy rate in the era of CT: an 18-year perspective. Radiology. 2010 Aug;256(2):460-5. doi: 10.1148/radiol.10091570. Epub 2010 Jun 7. PMID 20529988
- [Background] Rogers W, Hoffman J, Noori N. Harms of CT scanning prior to surgery for suspected appendicitis. Evid Based Med. 2015 Feb;20(1):3-4. doi: 10.1136/ebmed-2014-110075. Epub 2014 Nov 27. PMID 25429870
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Background] Lynge E, Sandegaard JL, Rebolj M. The Danish National Patient Register. Scand J Public Health. 2011 Jul;39(7 Suppl):30-3. doi: 10.1177/1403494811401482. PMID 21775347
- [Background] Pedersen CB. The Danish Civil Registration System. Scand J Public Health. 2011 Jul;39(7 Suppl):22-5. doi: 10.1177/1403494810387965. PMID 21775345
- [Background] Kleif J, Thygesen LC, Gogenur I. Validity of the diagnosis of appendicitis in the Danish National Patient Register. Scand J Public Health. 2020 Feb;48(1):38-42. doi: 10.1177/1403494818761765. Epub 2018 Mar 19. PMID 29554842
- [Background] Sallinen V, Akl EA, You JJ, Agarwal A, Shoucair S, Vandvik PO, Agoritsas T, Heels-Ansdell D, Guyatt GH, Tikkinen KA. Meta-analysis of antibiotics versus appendicectomy for non-perforated acute appendicitis. Br J Surg. 2016 May;103(6):656-667. doi: 10.1002/bjs.10147. Epub 2016 Mar 17. PMID 26990957
- See also: Protocol — https://drive.google.com/file/d/1W54pSz_HHao0iGrteYMsJyCADH5aQnYL/view?usp=sharing